CLINICAL TRIAL: NCT04621331
Title: An Open-label, Multicenter Study Investigating the Efficacy, Safety and Pharmacokinetics of Roxadustat (FG-4592) for Treatment of Anemia in Pediatric Patients With Chronic Kidney Disease
Brief Title: Investigating the Efficacy, Safety and PK of Roxadustat (FG-4592) for Treatment of Anemia in Pediatric Patients With CKD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Kyntra Bio (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGN-PED-CLIN-02
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Anemia Associated With Chronic Kidney Disease
Keywords: Anemia, Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Roxadustat (Experimental): Starting doses of 20, 50, 70 or 100 mg based on weight.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — HIF-PH inhibitor for treatment of anemia in CKD
  Other Names: FG-4592

SUMMARY:
This open-labeled, multicenter study is designed to evaluate the efficacy, safety and PK/PD of roxadustat in ESA-naïve and ESA-treated pediatric patients with CKD Stages 3, 4, and 5, as well as end-stage renal disease (ESRD) who are receiving either hemodialysis (HD) or peritoneal dialysis (PD). The study will enroll patients between the ages of 2 to <18 years in two sequential cohorts, with the older cohort of ages 12 to <18 years enrolled first. Approximately 30 patients will be enrolled in each age-based cohort.

ELIGIBILITY:
Important Inclusion Criteria:

* Clinically stable CKD in the opinion of the investigator.
* Estimated glomerular filtration rate (Bedside Schwartz formula) of < 60 ml/min/1.73 m2 (stage 3, 4 and 5 CKD) for non-dialysis patients, or patients who are receiving chronic dialysis (hemodialysis or peritoneal dialysis) for ESRD.
* For ESA-naïve patients (either NDD or DD; ESA-naïve is defined as those patients whose total duration of prior ESA exposure is ≤ 3 weeks within the preceding 12 weeks at the time informed consent is obtained), mean of two most recent central laboratory Hb values during the screening period obtained at least 2 days apart must be < 11.0 g/dL. For patients currently receiving stable ESA dosing who will discontinue ESA and convert to roxadustat during study, mean of two most recent central laboratory Hb values during the screening period obtained at least 2 days apart must be ≥ 10.0 g/dL and ≤ 12.5 g/dL.
* Ferritin >50 ng/mL and transferrin saturation >10% (obtained from screening visit).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2x upper limit of normal (ULN) and total bilirubin (Tbili) ≤1.5x ULN at randomization (obtained from screening visit).
* Serum folate and vitamin B12 > LLN (obtained from screening visit).

Important Exclusion Criteria:

* Uncontrolled hypertension as judged by the principal investigator in the 2 weeks prior to screening.
* Known hematologic disease other than anemia associated with CKD.
* Known malignancy within the past 5 years before screening.
* Any prior organ transplant or any planned organ transplant during the study period.
* Any RBC transfusion during the past 8 weeks before screening.
* Any condition leading to significant blood loss (e.g., gastrointestinal bleeding, surgical procedures) within 8 weeks before screening or during the screening period.
* History of chronic liver disease.
* Pure red cell aplasia (PRCA) or history of PRCA.
* History of epileptic seizures.
* History of hyperlipidemia or significant thrombotic/thromboembolic event (e.g., deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction).
* History of thrombosis of an arteriovenous fistula/graft within 12 weeks prior to enrollment.
* Any active systemic or significant infection or episode of peritonitis within 30 days of screening.
* Any statin use within 30 days of screening.
* Any prior exposure to roxadustat or any other HIF-PH inhibitor.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with mean Hb ≥ 11.0 g/dL | Averaged over weeks 16-24

SECONDARY OUTCOMES:
Mean change in Hb | Baseline to averaged over weeks 16-24
Time to first Hb response (this only applies to NDD patients) | From baseline without rescue therapy

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Mount Sinai Hospital (MSH), New York, New York
  - Investigative site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No